CLINICAL TRIAL: NCT04001335
Title: Diagnosis of Cutaneous Leishmaniasis Using the CL-detect Rapid Test in Travelers and Migrants in Belgium
Acronym: RapidLeish
Status: Terminated | Type: Observational
Why Stopped: No patient recruitment possible during COVID-19, inavailability RDTs
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: 1298/19
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Cutaneous Leishmaniases
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CL suspicion: Patients with skin lesions suspected to be cutaneous leishmaniasis
  Interventions: Diagnostic Test: Dental Broach

INTERVENTIONS:
Diagnostic Test: Dental Broach — Dental broach, RDT and PCR

SUMMARY:
Cutaneous Leishmaniasis (CL) is a neglected tropical disease which is increasingly seen in travelers and migrants evaluated in travel clinics of non-endemic countries. Various CL species are present in different parts of the world, and these different species vary in severity, prognosis and therapeutic approaches.

At ITM, diagnosis of CL in suspected patients is done using a skin biopsy, analyzed by diagnostic PCR, and species typing PCR. This method is invasive, and diagnosis is often delayed for days to weeks.

The new antigen-based CL Detect Rapid Test uses dental broach sampling and has results within 30 minutes. Dental broach samples left over from the Cl Detect Rapid test may still be used for PCR including species typing.

How well the CL Detect Rapid Test performs in the varied population of a travel clinic and whether it is possible to use dental broach sampling for further PCR tests in this population needs to be evaluated The aim of this study is to study the performance of the CL Detect Rapid Test and whether dental broach sampling can replace skin biopsy for CL at ITM.

ELIGIBILITY:
Inclusion Criteria:

* Skin biopsy for leishmania test requested by treating ITM clinician OR
* externally requested skin biopsy for Leishmania tested at ITM with an ITM consultation <7 days of the biopsy sample
* willing and able to provide consent/assent
* not on CL treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspicion of CL will be screened for inclusion.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CL detect RDT | 2019-2010
  Against combined reference of microscopy and PCR using skin punch biopsy

SECONDARY OUTCOMES:
Proportion of PCR positives on dental broach sample | 2019-2020
  Compared to PCR positives on skin punch biopsy
Proportion of successful species typing on dental broach sample | 2019-2020
  Compared to successful species typing on skin punch biopsy sample

CONTACTS AND LOCATIONS:
Overall Officials: Saskia van Henten, MD, Principal Investigator — Institute of Tropical Medicine; Johan van Griensven, MD,PhD, Study Director — Institute of Tropical Medicine
Locations (1):
- Institute of Tropical Medicine, Antwerp, Belgium